CLINICAL TRIAL: NCT02666898
Title: Phase II, Multicenter, Trial, Exploring "Chemo-free" Treatment (GA101+Ibrutinib) and MRD-driven Strategy in Previously Untreated Symptomatic B-chronic Lymphocytic Leukemia Medically Fit. A FILO Study. A Study From the Goelams/GCFLLC/MW Intergroup
Brief Title: Phase II Trial GA101 Inbrutinib B CLL
Acronym: ICLL07GAI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Roche Pharma AG (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICLL07GAI
Record Dates: First submitted 2015-10-26; First posted 2016-01-28 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: Residual disease
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasm, Residual | interventions — obinutuzumab; ibrutinib; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Obinutuzumab and Ibrutinib CLL treatment (Experimental): 3 parts
  PART 1: 6 cycles of GA101 + Ibrutinib 420mg PO/ 28 days:
  GA101:
  C 1 D1: 100mg, D2: 900mg D8 and D15: 1000 mg i.v C 2 to 6 :D1 1000 mg i.v
  Ibrutinib:
  D3 Month 1 to Day 30 Month 15: 420mg daily PO
  PART 2: 4 cycles / 28 days
  After evaluation at D1 month 9:
  * patients in CR with BM MRD < 10-4, Ibrutinib 420mg daily
  * patients with BM MRD >10-4 or PR 4 courses of GA101 + FC/ 28-day + Ibrutinib PO until M16 Cycle 1 to 4 - GA101: 1000 mg i.v on day 1
  * Fludarabine : 40 mg/m² per os, days 2-4, / 28 days
  * Cyclophosphamide : 250 mg/m² per os, days 2-4, / 28 days
  * Ibrutinib 420mg/day PO
  PART 3 (only in GAI-FC+Ibru arm) :
  After evaluation at D1 of M16:
  * patients CR with BM MRD< 10-4, treatment stopped
  * patients CR with BM MRD >10-4, Ibrutinib continued until PD or PB MRD becomes negative.
  Interventions: Drug: GA101; Drug: Ibrutinib; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: GA101 — Part 1 :6 cycles
  Obinutuzumab/GA101:
  First cycle:
  D1: 100mg, D2: 900mg D8 and D15: 1000 mg i.v
  Cycle 2 to 6 (every 28 days) :
  D1 of every cycle: 1000 mg i.v PART 2 4 cycles
  -patients have BM MRD >10-4 or PR: Cycle 1 to 4 Obitinuzumab/GA101: 1000 mg i.v on day 1
  Other Names: Obinutuzumab
Drug: Ibrutinib — Part 1 :6 cycles
  Cycle 2 to 6 (every 28 days) :Ibrutinib:
  D3 Month 1 to Day 30 Month 15: 420mg daily PO PART 2:4 cycles
  * patients in CR with BM MRD < 10-4 : Ibrutinib alone 420mg daily
  * patients with BM MRD >10-4 whatever responses or PR :Cycle 1 to 4 Ibrutinib 420mg daily with Cyclophosphamide and Fludarabine
  Other Names: Imbruvica
Drug: Cyclophosphamide — PART 2 :
  patients with BM MRD >10-4 or PR (except PD and SD), receive : 4 cycles of FC+GA101 every 28 days Cyclophosphamide : 250 mg/m² per os, D2 to D4 in association with GA101, ibrutinib and fludarabine
  Other Names: Endoxan
Drug: Fludarabine — PART 2 :
  patients with BM MRD >10-4 or PR (except PD and SD), receive : 4 cycles of FC+GA101 every 28 days : Fludarabine : 40 mg/m² per os, D2 to D4 in association with GA101, ibrutinib and cyclophosphamide
  Other Names: Fludara

SUMMARY:
Phase II study testing chemo-free induction therapy with Ibrutinib + Obinutuzumab nine months /

Study Part 1:

All patients will receive 8 courses of GA101 + ibrutinib 420mg PO every 28 days

Study Part 2:

After evaluation at D1 of month 9:

If patients are in CR with BM MRD < 10-4, they will continue ibrutinib alone at a dose of 420mg daily If patients have BM MRD >10-4 whatever IWCLL 2008 responses or PR they will receive four courses of GA101 + FC at 28-day intervals + Ibrutinib PO until final evaluation of M16

DETAILED DESCRIPTION:
Phase II study testing chemo-free induction therapy with Ibrutinib + Obinutuzumab during nine months followed by a MRD-driven strategy. Assessment of response as well as bone marrow MRD evaluation will be performed at Day 1 month 9:

1. Patients reaching CR with marrow MRD below 10-4 threshold will continue ibrutinib during 6 additional months.
2. Patients in PR or bone marrow MRD > 10-4 will receive Ibrutinib during 6 additional months and 4 courses of FC+ GA101. At Day 1 Month 16, patients in CR but with MRD> 10-4 will continue Ibrutinib until progressive disease.
3. Patients in stable or progressive disease will be excluded out of the trial.

Final evaluation of response (with BM MRD) will be performed at Day 1 Month 16.

ELIGIBILITY:
Inclusion Criteria:

* Patient information and written informed consent
* Age 18 years or older
* Immunophenotypically confirmed B-CLL (IWCLL2008 and Matutes score 4 or 5)
* Binet stage C according to IWCLL 2008 criteria or Binet stage A and B with active disease could be considered for inclusion.
* Patients with no prior treatment (chemotherapy, radiotherapy, immunotherapy) except steroids for less than 1 month
* Absence of 17p deletion as assessed by FISH (< 10 % positive nuclei)
* Performance status ECOG < 2
* CIRS (Cumulative Illness Rating Scale) ≤ 6 (see appendix 4 for calculation of CIRS score) Mandatory inclusion criteria for treatment with ibrutinib

Hematology values must be within the following limits:

* Absolute neutrophil count (ANC) <1 G/L independent of growth factor support
* Platelets <100 G/L or <50 G/L if bone marrow involvement independent of transfusion support in either situation

Biochemical values within the following limits:

* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Serum creatinine ≤ 2 x ULN or estimated Glomerular Filtration Rate (Cockroft Gault≥ 40 mL/min/1.73m2
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [Beta-hCG]) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study, including biomarkers, and are willing to participate in the study

Exclusion Criteria:

* Binet stage A and B without active disease according to IWCLL 2008 criteria

  * Known HIV seropositivity
  * Hepatitis B or C seropositivity (unless clearly due to vaccination)
  * Active hemolysis (isolated positive DAT is not an exclusion criteria)
  * Life expectancy < 6 months
  * Patient refusal to perform the bone marrow biopsy for evaluation points
  * Clinically significant auto-immune anemia
  * Active second malignancy currently requiring treatment (except basal cell carcinoma in situ endometrial carcinoma and incidental prostate carcinoma) and/or less than 5 years CR after breast cancer
  * Any severe co-morbid conditions such as Class III or IV heart failure, myocardial infarction within months, unstable angina, ventricular tachyarrhythmias requiring ongoing treatment, severe chronic obstructive pulmonary disease with hypoxemia, uncontrolled diabetes mellitus, or uncontrolled hypertension
  * Concomitant disease requiring prolonged use of corticosteroids (> 1 month)
  * Known hypersensitivity with anaphylactic reaction to humanized monoclonal antibodies or any of the study drugs
  * Contraindication to the use of Obinutuzumab.
  * Contraindication to use of Ibrutinib
  * Transformation to aggressive B-cell malignancy (e.g. diffuse large cell lymphoma, Hodgkin lymphoma, or prolymphocytic leukaemia)
  * Active bacterial, viral or fungal infection
  * Abnormal renal function with creatinine clearance < 60 ml/min calculated according to the formula of Cockcroft and Gault
  * Total bilirubin, gamma glutamyltransferase or transaminase levels > 2.5 ULN.
  * Any coexisting medical or psychological condition that would preclude participation in the required study procedures
  * Patient with mental deficiency preventing proper understanding of the requirements of treatment.
  * Pregnant or breastfeeding women.
  * Adult under law-control
  * Fertile male and female patients who cannot or do not wish to use an effective method of contraception, during and for 18 months after the final treatment used for the purposes of the study.
  * No affiliate to social security

Mandatory exclusion criteria for treatment with Ibrutinib

* Major surgery within 4 weeks of randomization.
* Known central nervous system lymphoma.
* History of stroke or intracranial hemorrhage within 6 months prior to randomization.
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong CYP3A inhibitors.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
* Known history of human immunodeficiency virus (HIV) or active Hepatitis C Virus or active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics.
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
Study treatment response | month 16
  IWCLL criteria response
Study treatment response | month 16
  MRD

SECONDARY OUTCOMES:
progression free survival | month 16
  relapse
progression free survival | month 16
  death
overall survival | month 16
  death
time to next treatment | 36 months
  date of new treatment after first relapse

CONTACTS AND LOCATIONS:
Overall Officials: Valérie ROUILLE, Mrs, Study Director — French Innovative Leukemia Organisation; Pierre FEUGIER, MD PD, Principal Investigator — French Innovative Leukemia Organisation; Anne Sophie MICHALLET, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Sponsor FILO, Tours, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Michallet AS, Letestu R, Le Garff-Tavernier M, Campos L, Ticchioni M, Dilhuydy MS, Morisset S, Rouille V, Mahe B, Laribi K, Villemagne B, Ferrant E, Tournilhac O, Delmer A, Molina L, Leblond V, Tomowiak C, de Guibert S, Orsini-Piocelle F, Banos A, Carassou P, Cartron G, Fornecker LM, Ysebaert L, Dartigeas C, Truchan-Graczyk M, Vilque JP, Schleinitz TA, Cymbalista F, Lepretre S, Levy V, Nguyen-Khac F, Feugier P. A fixed-duration immunochemotherapy approach in CLL: 5.5-year results from the phase 2 ICLL-07 FILO trial. Blood Adv. 2023 Aug 8;7(15):3936-3945. doi: 10.1182/bloodadvances.2022009594. PMID 37026799
- [Derived] Michallet AS, Letestu R, Le Garff-Tavernier M, Aanei C, Ticchioni M, Dilhuydy MS, Subtil F, Rouille V, Mahe B, Laribi K, Villemagne B, Salles G, Tournilhac O, Delmer A, Portois C, Pegourie B, Leblond V, Tomowiak C, De Guibert S, Orsini Piocelle F, Banos A, Carassou P, Cartron G, Fornecker LM, Ysebaert L, Dartigeas C, Truchan-Graczyk M, Vilque JP, Aurran T, Cymbalista F, Lepretre S, Levy V, Nguyen-Khac F, Feugier P. A fixed-duration, measurable residual disease-guided approach in CLL: follow-up data from the phase 2 ICLL-07 FILO trial. Blood. 2021 Feb 25;137(8):1019-1023. doi: 10.1182/blood.2020008164. PMID 33167024
- [Derived] Michallet AS, Dilhuydy MS, Subtil F, Rouille V, Mahe B, Laribi K, Villemagne B, Salles G, Tournilhac O, Delmer A, Portois C, Pegourie B, Leblond V, Tomowiak C, de Guibert S, Orsini F, Banos A, Carassou P, Cartron G, Fornecker LM, Ysebaert L, Dartigeas C, Truchan Graczyk M, Vilque JP, Aurran T, Cymbalista F, Lepretre S, Levy V, Nguyen-Khac F, Le Garff-Tavernier M, Aanei C, Ticchioni M, Letestu R, Feugier P. Obinutuzumab and ibrutinib induction therapy followed by a minimal residual disease-driven strategy in patients with chronic lymphocytic leukaemia (ICLL07 FILO): a single-arm, multicentre, phase 2 trial. Lancet Haematol. 2019 Sep;6(9):e470-e479. doi: 10.1016/S2352-3026(19)30113-9. Epub 2019 Jul 16. PMID 31324600
- See also: FILO internet site — http://www.filo-leucemie.org